CLINICAL TRIAL: NCT01718860
Title: Effects of Postoperative Residual Paralysis on Costs of Hospital Care, Length of Hospitalization and Intensive Care Unit Admission Rate
Brief Title: Effects of Postoperative Residual Paralysis on Hospital Costs
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Matthias Eikermann, Dr., Massachusetts General Hospital
Other Study IDs: 2016P002695; IISP#39443 (Other Grant/Funding Number: MERCK & CO INC)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Residual Paralysis, Post-Anesthesia
Keywords: Cost Analysis; Postoperative Complications; Length of Stay; Intensive Care Units
MeSH Terms: conditions — Delayed Emergence from Anesthesia; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Postoperative Residual Paralysis: Patients with train-of-four ratio less than 0.9 measured in the postanesthesia care unit
  Interventions: Procedure: Quantitative measurement of neuromuscular transmission
- No Postoperative Residual Paralysis: Patients with train-of-four ratio greater than 0.9 measured in the postanesthesia care unit
  Interventions: Procedure: Quantitative measurement of neuromuscular transmission

INTERVENTIONS:
Procedure: Quantitative measurement of neuromuscular transmission — Quantitative measurement of neuromuscular transmission with train-of-four watches.

SUMMARY:
This is a secondary analysis of a previously performed prospective, observer-blinded, observational study at Massachusetts General Hospital. The primary aim of this study is to evaluate the effects of residual paralysis at admission to the post-anesthesia care unit (PACU) on total costs of hospital care.

Secondary analyses will be conducted to evaluate the effects of postoperative residual paralysis on potential cost-influencing factors, i.e. incidence of minor and major postoperative respiratory complications, hospital length of stay (LOS), unplanned intensive care unit (ICU) admission rate, as well as length of stay in the PACU.

ELIGIBILITY:
Inclusion Criteria:

* Each subject has been given non-depolarizing neuromuscular blocking agents as part of general anesthesia.
* Each subject must be at least 18 years of age
* Train-of-four monitoring in the post-anesthesia care unit

Exclusion Criteria:

* The subject is scheduled to be transferred to an intensive care unit after surgery.
* Children and pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who arrived at the post-anesthesia care unit after receiving neuromuscular blocking agents as part of their surgical anaesthesia.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Hospital costs | Patients will be followed from date of admission to date of hospital discharge, an expected 2 days to 4 weeks

SECONDARY OUTCOMES:
Hospital Length of Stay | within 100 days after surgery

OTHER OUTCOMES:
Incidence of postoperative respiratory complications | Within one month after surgery
Incidence of unplanned postoperative intensive care unit admission | Within one week after surgery
  Incidence of unplanned postoperative intensive care unit admission due to respiratory failure, pulmonary edema and arrhythmia.
Length of stay in the post-anesthesia care unit (PACU) | Patients will be followed until PACU discharge, an expected 2 days to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD, PhD, Principal Investigator — Partners
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Butterly A, Bittner EA, George E, Sandberg WS, Eikermann M, Schmidt U. Postoperative residual curarization from intermediate-acting neuromuscular blocking agents delays recovery room discharge. Br J Anaesth. 2010 Sep;105(3):304-9. doi: 10.1093/bja/aeq157. Epub 2010 Jun 24. PMID 20576632
- [Background] Herbstreit F, Zigrahn D, Ochterbeck C, Peters J, Eikermann M. Neostigmine/glycopyrrolate administered after recovery from neuromuscular block increases upper airway collapsibility by decreasing genioglossus muscle activity in response to negative pharyngeal pressure. Anesthesiology. 2010 Dec;113(6):1280-8. doi: 10.1097/ALN.0b013e3181f70f3d. PMID 20980910
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Background] Berg H, Roed J, Viby-Mogensen J, Mortensen CR, Engbaek J, Skovgaard LT, Krintel JJ. Residual neuromuscular block is a risk factor for postoperative pulmonary complications. A prospective, randomised, and blinded study of postoperative pulmonary complications after atracurium, vecuronium and pancuronium. Acta Anaesthesiol Scand. 1997 Oct;41(9):1095-1103. doi: 10.1111/j.1399-6576.1997.tb04851.x. PMID 9366929
- [Background] Grosse-Sundrup M, Henneman JP, Sandberg WS, Bateman BT, Uribe JV, Nguyen NT, Ehrenfeld JM, Martinez EA, Kurth T, Eikermann M. Intermediate acting non-depolarizing neuromuscular blocking agents and risk of postoperative respiratory complications: prospective propensity score matched cohort study. BMJ. 2012 Oct 15;345:e6329. doi: 10.1136/bmj.e6329. PMID 23077290
- [Background] Sasaki N, Meyer MJ, Malviya SA, Stanislaus AB, MacDonald T, Doran ME, Igumenshcheva A, Hoang AH, Eikermann M. Effects of neostigmine reversal of nondepolarizing neuromuscular blocking agents on postoperative respiratory outcomes: a prospective study. Anesthesiology. 2014 Nov;121(5):959-68. doi: 10.1097/ALN.0000000000000440. PMID 25225821
- [Derived] Grabitz SD, Rajaratnam N, Chhagani K, Thevathasan T, Teja BJ, Deng H, Eikermann M, Kelly BJ. The Effects of Postoperative Residual Neuromuscular Blockade on Hospital Costs and Intensive Care Unit Admission: A Population-Based Cohort Study. Anesth Analg. 2019 Jun;128(6):1129-1136. doi: 10.1213/ANE.0000000000004028. PMID 31094777